CLINICAL TRIAL: NCT06851091
Title: Investigation of the Relationship Between Central Sensitization Parameters and Balance Changes in Patients With Fibromyalgia
Brief Title: Investigation of the Relationship Between Central Sensitization and Balance in Fibromyalgia
Status: Recruiting | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Feyza Nur Yucel, Principal Investigator, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Other Study IDs: 24/759
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Fibromyalgia Syndrome; Central Sensitisation; Postural Balance
Keywords: Fibromyalgia; Central Sensitisation; Balance Changes; Postural Balance
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (Healthy volunteers): Healthy volunteers without a diagnosis of Fibromyalgia Syndrome will be included in Group 1. (n=20)
  Interventions: Diagnostic Test: Biodex Balance System; Diagnostic Test: Pressure Pain Threshold (PPT) Measurement with Algometer; Diagnostic Test: Conditioned Pain Modulation (CPM); Diagnostic Test: Slowly Repeated Evoked Pain Assessment Protocol (SREP); Diagnostic Test: Central Sensitization Inventory (CSI); Diagnostic Test: Numeric Rating Scale (NRS); Diagnostic Test: Revised Fibromyalgia Impact Questionnaire (FIQ); Diagnostic Test: S-LANSS Pain Score (Self-administered Leeds Assessment of Neuropathic Symptoms and Signs); Diagnostic Test: Tampa Kinesiophobia Scale (TKS); Diagnostic Test: Hospital Anxiety and Depression Scale (HAD); Diagnostic Test: SF-12 Health Survey (SF-12 Quality of Life Scale); Diagnostic Test: Fatigue Severity Scale (FSS); Diagnostic Test: Timed Up and Go Test (TUG)
- Group 2 (Patients with fibromyalgia syndrome): Patients diagnosed with Fibromyalgia Syndrome according to ACR 2016 criteria will be included in Group 2. (n=55)
  Interventions: Diagnostic Test: Biodex Balance System; Diagnostic Test: Pressure Pain Threshold (PPT) Measurement with Algometer; Diagnostic Test: Conditioned Pain Modulation (CPM); Diagnostic Test: Slowly Repeated Evoked Pain Assessment Protocol (SREP); Diagnostic Test: Central Sensitization Inventory (CSI); Diagnostic Test: Numeric Rating Scale (NRS); Diagnostic Test: Revised Fibromyalgia Impact Questionnaire (FIQ); Diagnostic Test: S-LANSS Pain Score (Self-administered Leeds Assessment of Neuropathic Symptoms and Signs); Diagnostic Test: Tampa Kinesiophobia Scale (TKS); Diagnostic Test: Hospital Anxiety and Depression Scale (HAD); Diagnostic Test: SF-12 Health Survey (SF-12 Quality of Life Scale); Diagnostic Test: Fatigue Severity Scale (FSS); Diagnostic Test: Timed Up and Go Test (TUG)

INTERVENTIONS:
Diagnostic Test: Biodex Balance System — Biodex Balance System [Biodex Balance System SD (Biodex, Inc, Shirley, NY) (BBS)]:The Biodex Balance System is a computer-assisted device that assesses postural stability. It measures static and dynamic balance, fall risk, and proprioception through different difficulty levels and test protocols. In our study, this system will be used to investigate the relationship between balance and central sensitization. Participants will be evaluated using the postural stability test, fall risk test, athlete single leg test, and limits of stability test protocols, and they will be trained before the testing process.
Diagnostic Test: Pressure Pain Threshold (PPT) Measurement with Algometer — Pressure pain threshold (PPT) is defined as the minimum force applied that causes pain. This measurement is commonly used for assessing tender points and has been shown to be useful.
Diagnostic Test: Conditioned Pain Modulation (CPM) — According to this protocol, a pressure stimulus, referred to as the test stimulus, will first be applied to the trapezius muscle to induce a pain intensity of 4 on a 10-point Numeric Rating Scale (NRS). Subsequently, a conditioning stimulus will be introduced by immersing the participant's right hand in 7°C water for 20 seconds. Following this conditioning stimulus, the same test stimulus will be reapplied to the trapezius muscle, and participants will be asked to rate their pain using the NRS. If participants are unable to keep their hands in the water for the full 20 seconds, the test stimulus will be applied immediately after hand removal. The CPM score will be calculated as the ratio of the initial NRS score to the second NRS score, multiplied by 100. Scores above 100 are considered indicative of a normal CPM response, with higher scores reflecting greater descending pain inhibition.
Diagnostic Test: Slowly Repeated Evoked Pain Assessment Protocol (SREP) — Responses to induced pain indicate the presence of allodynia and hyperalgesia in FMS patients. The Slow Repetitive Evoked Pain (SREP) protocol consists of nine suprathreshold painful stimuli applied to the nail bed for five seconds each, with 30-second intervals. Painful stimulation will be administered using a pressure algometer with a 1 cm² stimulation surface. Nailbed pain stimuli are commonly used to assess pain sensitivity.
  The intensity of pain perception from each SREP stimulus will be evaluated using a 10-point Numerical Rating Scale (NRS) (0 = no pain, 10 = extremely painful). The SREP sensitization index will be calculated as the difference between the final and initial pain scores.
  Higher positive SREP sensitization index values indicate a greater increase in perceived pain intensity across the nine stimuli, reflecting higher pain sensitization.
Diagnostic Test: Central Sensitization Inventory (CSI) — The Central Sensitization Inventory (CSI) is used by some researchers to investigate pain sensitivity through symptoms associated with central sensitization and related comorbidities. It can help determine the severity of central sensitization.
  The scale was developed to detect central sensitization in patients with chronic pain and consists of two sections: Section A and Section B. For scoring purposes, only Section A is used. A score of 40 or higher out of 100 is associated with an increased likelihood of central sensitization.
  This scale has been shown to be a reliable and valid tool in the Turkish population with chronic pain (test-retest reliability = 0.92, Cronbach's alpha = 0.93)
Diagnostic Test: Numeric Rating Scale (NRS) — Numeric Rating Scale (NRS) will be used to determine pain intensity during assessments. Participants will be asked to rate their pain intensity by selecting a value between 0 and 10. Higher scores are associated with increased pain severity.
Diagnostic Test: Revised Fibromyalgia Impact Questionnaire (FIQ) — Revised Fibromyalgia Impact Questionnaire (FIQ) consists of three sections: function, general, and symptoms, with a total of 21 questions. It evaluates the limitations and functional disability that occur in patients with fibromyalgia. All questions are scored on the Numeric Rating Scale (NRS), ranging from 0 to 10. As the score from the questionnaire increases, it indicates a higher level of disability related to fibromyalgia. In our study, the Turkish version of the questionnaire, which has been validated and shown to be reliable, will be used.
Diagnostic Test: S-LANSS Pain Score (Self-administered Leeds Assessment of Neuropathic Symptoms and Signs) — The S-LANSS pain score is a 7-item self-administered scale developed and validated to recognize neuropathic pain in chronic pain patients and distinguish it from nociceptive pain. It evaluates neuropathic symptoms and signs through a series of questions that help identify features like hyperalgesia, allodynia, and paresthesia, which characterize the chronic pain sensation associated with neuropathic pain. These features are often seen in fibromyalgia (FMS) pain. In our study, the Turkish version of the questionnaire, which has undergone validity and reliability testing, will be used.
Diagnostic Test: Tampa Kinesiophobia Scale (TKS) — The Tampa Kinesiophobia Scale is a 17-item measure designed to assess fear of movement/re-injury. The scale evaluates fear-avoidance behaviors related to work activities, injury/re-injury concerns, and fear-avoidance parameters. It is used in the context of acute and chronic low back pain, fibromyalgia (FMS), musculoskeletal injuries, and whiplash-associated disorders.
  The scale uses a 4-point Likert scoring system (1 = Strongly disagree, 4 = Strongly agree). After reversing the scores for items 4, 8, 12, and 16 (for example, if a participant selects 1 for these items, it is counted as 4; 2 is counted as 3, etc.), the total score is calculated. The participant receives a score between 17 and 68. A higher score on the scale indicates a higher level of kinesiophobia. In our study, the Turkish version of the scale, which has undergone validity and reliability testing, will be used.
Diagnostic Test: Hospital Anxiety and Depression Scale (HAD) — This scale is used to assess anxiety and depression symptoms and consists of 14 items (7 items for anxiety, 7 items for depression). For each subscale, scores range from 0 to 21:
  * 0-7 points: No symptoms or very mild symptoms
  * 8-10 points: Moderate symptoms
  * 11 points or higher: Symptoms likely corresponding to a clinical diagnosis of anxiety and depression According to the 2016 diagnostic criteria for Fibromyalgia Syndrome (FMS), the presence of depression contributes to the diagnosis of FMS. The HAD scale has been shown to be a suitable tool for assessing FMS and related patient education programs.
  In our study, the Turkish version of the HAD scale, which has been validated and shown to be reliable, will be used.
Diagnostic Test: SF-12 Health Survey (SF-12 Quality of Life Scale) — The SF-12 Health Survey is one of the most widely used scales for assessing health-related quality of life. In our study, the Turkish version of the SF-12, which has been validated and shown to be reliable, will be used. The scores will be calculated using an online calculation tool, and two types of scores-Physical Component Summary (PCS) and Mental Component Summary (MCS)-will be obtained.
Diagnostic Test: Fatigue Severity Scale (FSS) — The Fatigue Severity Scale (FSS) is a 9-item questionnaire used to assess the severity, frequency, and impact of fatigue on daily life. Each item is rated on a scale from 1 to 7. A lower score indicates a decrease in fatigue severity. In our study, the Turkish version of the scale, which has been validated and shown to be reliable, will be used.
Diagnostic Test: Timed Up and Go Test (TUG) — The Timed Up and Go (TUG) test is designed to measure dynamic balance based on the time it takes for participants to stand up and walk. The patient begins by sitting on a standardized chair (height of 46 cm). During the test, the patient is asked to stand up from the chair, walk 3 meters, turn around, and return to sit back on the chair. The time taken to complete this process is measured. Lower values indicate better stability. A cut-off value of 13.5 seconds is used to identify individuals at higher risk of falling.

SUMMARY:
The aim of the study is to investigate the relationship between central sensitization parameters and changes in static and dynamic balance in patients with fibromyalgia.

The main questions it aims to answer are:

* Do central sensitization parameters differ in patients with fibromyalgia compared to healthy individuals?
* How is balance performance in these individuals compared to healthy controls?
* Do central sensitization parameters affect static and dynamic balance in patients with fibromyalgia?
* Do central sensitization parameters lead to quantitative changes in balance in patients with fibromyalgia?

DETAILED DESCRIPTION:
Fibromyalgia is a syndrome characterized by chronic and widespread musculoskeletal pain. It is often accompanied by other symptoms such as fatigue, bowel disorders, sleep disturbances, and mood changes. It is estimated that fibromyalgia syndrome (FMS) affects approximately 2% to 8% of the global population.

The American College of Rheumatology (ACR) diagnostic criteria, based on the presence of multiple tender points, widespread chronic pain, somatic symptoms (such as headaches and abdominal pain), and cognitive symptoms, are used to diagnose individuals with fibromyalgia syndrome (FMS). Widespread pain, headaches, muscle spasms, and balance disorders are the most common symptoms leading to physical disability. These disabling symptoms reduce quality of life and make daily activities more difficult. The impact of these symptoms results in an annual cost of €7,256-7,900 per diagnosed patient in developed countries, creating a secondary socioeconomic burden . This burden includes high absenteeism, unemployment, early retirement, and an increased number of sick leave days.

Postural stability is a complex task required to maintain balance and orientation in a gravity-based environment. This task necessitates the rapid and dynamic integration of sensory information from the somatosensory, vestibular, and visual systems, which are essential for maintaining balance. Changes in balance are associated with poor balance confidence, which increases the risk of falls. Balance disorders are among the most common symptoms in patients with fibromyalgia syndrome (FMS), with a prevalence ranging from 45% to 68%. Previous studies have demonstrated that balance disorders are more prevalent in FMS patients compared to healthy individuals. Furthermore, in FMS patients with impaired balance, a correlation has been shown between balance disorders and an increased risk and/or frequency of falls. However, the underlying mechanism of balance problems in these patients has not yet been elucidated.

FMS is known to originate from a central sensitization phenomenon. According to the International Association for the Study of Pain, central sensitization is defined as an increased response of central nervous system (CNS) neurons to normal or subthreshold afferent inputs. It is hypothesized that changes in postural control may be a response to impaired sensory processing within the CNS and that the increased responsiveness of nociceptive neurons and the presence of central sensitization in the CNS may affect postural control processing, altering neuromuscular interactions and disrupting balance.

Central sensitization, one of the key mechanisms in the pathogenesis of FMS, has been reported to play a significant role in balance control in a study conducted by Sennholz et al. on patients with migraines. In this study, which included migraine patients and healthy controls, balance assessment was performed alongside an evaluation of central sensitization using quantitative sensory tests (cold and heat pain thresholds, mechanical pain thresholds, and pressure pain thresholds) and the central sensitization inventory. The results demonstrated that balance impairment in migraine patients was associated with a decreased pain threshold and an increased central sensitization inventory score.

To our knowledge, no study has yet quantitatively investigated the relationship between central sensitization levels and balance performance in FMS. Based on these findings, we aim to determine the relationship between central sensitization parameters and static and dynamic balance changes in FMS, a member of the central sensitivity syndrome family, similar to migraines. Furthermore, we seek to highlight the importance of future rehabilitation interventions targeting this relationship, thereby contributing to the existing literature.

The study will be conducted as an observational, single-center study at the Physical Medicine and Rehabilitation Clinic of Health Sciences University Sultan 2.Abdülhamid Han Training and Research Hospital, involving patients diagnosed with FMS and healthy volunteers.

As part of the study, demographic data including participants' age, gender, height, weight, body mass index, smoking and alcohol use, marital status, occupation, education level, current medications, presence of comorbidities, and duration of FMS diagnosis will be recorded. Patients will be evaluated once, and the assessment will consist of the following:

* Biodex Balance System [Biodex Balance System SD (Biodex, Inc, Shirley, NY) (BBS)]
* Quantitative Sensory Testing, including Pressure Pain Threshold Measurement with an Algometer and Conditioned Pain Modulation
* Slowly Repeated Evoked Pain Assessment Protocol
* Central Sensitization Inventory
* Numeric Rating Scale
* Revised Fibromyalgia Impact Questionnaire
* S-LANSS Pain Score
* Tampa Kinesiophobia Scale
* Hospital Anxiety and Depression Scale
* SF-12 Quality of Life Scale
* Fatigue Severity Scale
* Timed Up and Go Test

Number of Patients to be Included in the Study:The number of patients to be included in the study has been planned based on the study by Sennholz et al., published in May 2024, using G-power version 3.1. The study will include 20 healthy controls and 55 fibromyalgia patients.

Statistical Methods:The distribution pattern of the data and the tests to be applied will be determined based on the Kolmogorov-Smirnov test, skewness, and kurtosis values. If the data follow a parametric distribution, they will be presented as mean ± standard deviation and 95% confidence interval; if the data follow a non-parametric distribution, they will be presented as median ± interquartile range (IQR).

Pressure pain threshold measurements with the algometer, conditioned pain modulation measurements, slowly repeated evoked pain measurements, and balance parameters will be compared between the patient and control groups using independent group T-tests or Mann-Whitney U tests. The linear relationships between algometer pressure pain threshold measurements, conditioned pain modulation, slowly repeated evoked pain measurements, and clinical parameters will be examined using Spearman/Pearson correlation analysis. For parametric data, multiple regression models may be constructed based on the characteristics of the variables.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FMS according to the ACR 2016 diagnostic criteria
* Being between the ages of 18 and 65
* Being literate
* Providing informed consent by signing the voluntary consent form

Exclusion Criteria:

* Being under 18 years old or over 65 years old
* Presence of vestibular disorders
* Having undergone spinal and/or extremity surgery (such as for back/hip/knee/foot) within the last 6 months
* History of lower extremity amputation
* Presence of spinal deformities
* Peripheral arterial disease
* Vitamin B12 deficiency
* Any neurological disorder (e.g., stroke, traumatic brain injury, multiple sclerosis, Parkinson's disease, central nervous system malignancies, etc.)
* Severe cardiopulmonary insufficiency (stage 3-4)
* Uncontrolled systemic diseases such as hypertension and diabetes
* Presence of systemic inflammatory diseases, malignancies, or active infections
* Pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Fibromyalgia Syndrome according to ACR 2016 criteria
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-09-04 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pressure Pain Threshold (PPT) Measurement with Algometer | 5 months
  Pressure pain threshold (PPT) is defined as the minimum force applied that causes pain. This measurement is commonly used for assessing tender points and has been shown to be useful.
Conditioned Pain Modulation (CPM) | 5 months
  According to this protocol, a pressure stimulus, referred to as the test stimulus, will first be applied to the trapezius muscle to induce a pain intensity of 4 on a 10-point Numeric Rating Scale (NRS). Subsequently, a conditioning stimulus will be introduced by immersing the participant's right hand in 7°C water for 20 seconds. Following this conditioning stimulus, the same test stimulus will be reapplied to the trapezius muscle, and participants will be asked to rate their pain using the NRS. If participants are unable to keep their hands in the water for the full 20 seconds, the test stimulus will be applied immediately after hand removal. The CPM score will be calculated as the ratio of the initial NRS score to the second NRS score, multiplied by 100. Scores above 100 are considered indicative of a normal CPM response, with higher scores reflecting greater descending pain inhibition.
Slowly Repeated Evoked Pain Assessment Protocol (SREP) | 5 months
  Responses to induced pain indicate the presence of allodynia and hyperalgesia in FMS patients. The Slowly Repeated Evoked Pain Assessment Protocol (SREP) consists of nine suprathreshold painful stimuli applied to the nail bed for five seconds each, with 30-second intervals. Painful stimulation will be administered using a pressure algometer with a 1 cm² stimulation surface. Nailbed pain stimuli are commonly used to assess pain sensitivity. The intensity of pain perception from each SREP stimulus will be evaluated using a 10-point Numerical Rating Scale (NRS) (0 = no pain, 10 = extremely painful). The SREP sensitization index will be calculated as the difference between the final and initial pain scores. Higher positive SREP sensitization index values indicate a greater increase in perceived pain intensity across the nine stimuli, reflecting higher pain sensitization.

SECONDARY OUTCOMES:
Biodex Balance System | 5 months
  [Biodex Balance System SD (Biodex, Inc, Shirley, NY) (BBS)]:The Biodex Balance System is a computer-assisted device that assesses postural stability. It measures static and dynamic balance, fall risk, and proprioception through different difficulty levels and test protocols. In our study, this system will be used to investigate the relationship between balance and central sensitization. Participants will be evaluated using the postural stability test, fall risk test, athlete single leg test, and limits of stability test protocols, and they will be trained before the testing process.
The Central Sensitization Inventory (CSI) | 5 months
  The Central Sensitization Inventory (CSI) is used by some researchers to investigate pain sensitivity through symptoms associated with central sensitization and related comorbidities. It can help determine the severity of central sensitization. The scale was developed to detect central sensitization in patients with chronic pain and consists of two sections: Section A and Section B. For scoring purposes, only Section A is used. A score of 40 or higher out of 100 is associated with an increased likelihood of central sensitization. This scale has been shown to be a reliable and valid tool in the Turkish population with chronic pain (test-retest reliability = 0.92, Cronbach's alpha = 0.93)
Numeric Rating Scale (NRS) | 5 months
  Numeric Rating Scale (NRS) will be used to determine pain intensity during assessments. Participants will be asked to rate their pain intensity by selecting a value between 0 and 10. Higher scores are associated with increased pain severity.
Revised Fibromyalgia Impact Questionnaire (FIQ) | 5 months
  Revised Fibromyalgia Impact Questionnaire (FIQ) consists of three sections: function, general, and symptoms, with a total of 21 questions. It evaluates the limitations and functional disability that occur in patients with fibromyalgia. All questions are scored on the Numeric Rating Scale (NRS), ranging from 0 to 10. As the score from the questionnaire increases, it indicates a higher level of disability related to fibromyalgia. In our study, the Turkish version of the questionnaire, which has been validated and shown to be reliable, will be used.
S-LANSS Pain Score (Self-administered Leeds Assessment of Neuropathic Symptoms and Signs) | 5 months
  The S-LANSS pain score is a 7-item self-administered scale developed and validated to recognize neuropathic pain in chronic pain patients and distinguish it from nociceptive pain. It evaluates neuropathic symptoms and signs through a series of questions that help identify features like hyperalgesia, allodynia, and paresthesia, which characterize the chronic pain sensation associated with neuropathic pain. These features are often seen in fibromyalgia (FMS) pain. In our study, the Turkish version of the questionnaire, which has undergone validity and reliability testing, will be used.
Tampa Kinesiophobia Scale (TKS) | 5 months
  The Tampa Kinesiophobia Scale is a 17-item measure designed to assess fear of movement/re-injury. The scale evaluates fear-avoidance behaviors related to work activities, injury/re-injury concerns, and fear-avoidance parameters. It is used in the context of acute and chronic low back pain, fibromyalgia (FMS), musculoskeletal injuries, and whiplash-associated disorders. The scale uses a 4-point Likert scoring system (1 = Strongly disagree, 4 = Strongly agree). After reversing the scores for items 4, 8, 12, and 16 (for example, if a participant selects 1 for these items, it is counted as 4; 2 is counted as 3, etc.), the total score is calculated. The participant receives a score between 17 and 68. A higher score on the scale indicates a higher level of kinesiophobia. In our study, the Turkish version of the scale, which has undergone validity and reliability testing, will be used.
Hospital Anxiety and Depression Scale (HAD) | 5 months
  This scale is used to assess anxiety and depression symptoms and consists of 14 items (7 items for anxiety, 7 items for depression). For each subscale, scores range from 0 to 21:
  * 0-7 points: No symptoms or very mild symptoms
  * 8-10 points: Moderate symptoms
  * 11 points or higher: Symptoms likely corresponding to a clinical diagnosis of anxiety and depression According to the 2016 diagnostic criteria for Fibromyalgia Syndrome (FMS), the presence of depression contributes to the diagnosis of FMS. The HAD scale has been shown to be a suitable tool for assessing FMS and related patient education programs.
  In our study, the Turkish version of the HAD scale, which has been validated and shown to be reliable, will be used.
SF-12 Health Survey (SF-12 Quality of Life Scale) | 5 months
  The SF-12 Health Survey is one of the most widely used scales for assessing health-related quality of life. In our study, the Turkish version of the SF-12, which has been validated and shown to be reliable, will be used. The scores will be calculated using an online calculation tool, and two types of scores-Physical Component Summary (PCS) and Mental Component Summary (MCS)-will be obtained.
The Fatigue Severity Scale (FSS) | 5 months
  The Fatigue Severity Scale (FSS) is a 9-item questionnaire used to assess the severity, frequency, and impact of fatigue on daily life. Each item is rated on a scale from 1 to 7. A lower score indicates a decrease in fatigue severity. In our study, the Turkish version of the scale, which has been validated and shown to be reliable, will be used.
The Timed Up and Go (TUG) | 5 months
  The Timed Up and Go (TUG) test is designed to measure dynamic balance based on the time it takes for participants to stand up and walk. The patient begins by sitting on a standardized chair (height of 46 cm). During the test, the patient is asked to stand up from the chair, walk 3 meters, turn around, and return to sit back on the chair. The time taken to complete this process is measured. Lower values indicate better stability. A cut-off value of 13.5 seconds is used to identify individuals at higher risk of falling.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Ata, Asst. Prof., Study Director — Health Sciences University Sultan 2.Abdülhamid Han Training and Research Hospital; Feyza Nur Yücel, Specialist, Study Director — Health Sciences University Sultan 2.Abdülhamid Han Training and Research Hospital
Locations (1):
- Sultan 2. Abdülhamid Han Training and Research Hospital, İstanbul, Üsküdar, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Dataset sharing is not planned